CLINICAL TRIAL: NCT01847235
Title: The Efficacy and Safety of Temozolomide in Patients With Relapsed or Advanced Anaplastic Oligodendroglioma and Oligoastrocytoma: a Multicenter, Single-arm, Phase II Trial
Brief Title: Temozolomide in Relapsed or Advanced Anaplastic Oligodendroglioma and Oligoastrocytoma: Single-arm, Phase II Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Min Kim, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OD_OA
Record Dates: First submitted 2013-04-29; First posted 2013-05-06 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma
Keywords: Temozolomide
MeSH Terms: conditions — Oligodendroglioma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide (Experimental): Temozolomide 200 mg/m2/d in a fasting state for 5 consecutive days
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Temozolomide 200 mg/m2/d in a fasting state for 5 consecutive days (1,000 mg/m2 per 28-day cycle).
  Other Names: Temodal

SUMMARY:
The purpose of this study is to determine the efficacy and safety of temozolomide in patient with relapsed or advanced anaplastic oligodendroglioma and anaplastic oligoastrocytoma.

DETAILED DESCRIPTION:
Patient with relapsed or advanced anaplastic oligodendroglioma and anaplastic oligoastrocytoma will be enrolled. Enrolled patients will begin on temozolomide 200 mg/m2/d in a fasting state for 5 consecutive days (1,000 mg/m2 per 28-day cycle). Patients who were previously treated with any chemotherapy initially received temozolomide 150 mg/m2/d for 5 days (750 mg/m2 per cycle).Patients will be receving a total 6 cycles of chemotheray (4weeks/cycle * 6cycles = 24weeks). If the patients shows responses to Temozolomide, treatment can be continued by the investigator's discretion.

During the administration of Temozolomide, vital signs, physical examination, ECOG performance status, height, weight, hematology and chemistry test, adverse events and concomitant drugs will be evaluated every four weeks. Brain MRI for tumor assessment will be performed once every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven anaplastic oligodendroglioma or oligoastrocytoma
* Progressed or relapsed after surgery or radiation therapy
* Female or male aged 20 years or over
* At least 1 measurable mass lesion
* ECOG performance status 0-3
* Adequate organ function
* absolute neutrophil count > 1,500/μL
* platelet count > 75,000/μL
* hemoglobin greater than 9 g/dL or 900g/L
* serum creatinine less than 1.5 times the upper limit of laboratory normal
* total serum bilirubin less than 1.5 times the upper limit of laboratory normal
* AST or ALT less than three times the upper limit of laboratory normal

Exclusion Criteria:

* Prior course of temozolomide
* Combined glioblastoma
* Pregnant woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 6 month
  PFS will be examined with Kaplan-Meier method.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year
  ORR will be evaluated through the frequency analysis with 95% confidence interval.
Overall survival (OS) | 1 years
  OS will be examined with Kaplan-Meier method.
progression-free survival (PFS) | 1 year
  PFS will be examined with Kaplan-Meier method.
Number of Participants with Adverse Events | 1 years
  Regarding safety endpoints, all adverse events will be individually graded based on the CTCAE version 4.03. The number of participants with adverse events will be summarized using descriptive statistics.

OTHER OUTCOMES:
Predictive biomarker study | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tae Min Kim, MD, PhD, Study Chair — Seoul National University Hospital, Seoul, South Korea
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Perry JR, Rizek P, Cashman R, Morrison M, Morrison T. Temozolomide rechallenge in recurrent malignant glioma by using a continuous temozolomide schedule: the "rescue" approach. Cancer. 2008 Oct 15;113(8):2152-7. doi: 10.1002/cncr.23813. PMID 18756530
- [Background] Perry JR, Belanger K, Mason WP, Fulton D, Kavan P, Easaw J, Shields C, Kirby S, Macdonald DR, Eisenstat DD, Thiessen B, Forsyth P, Pouliot JF. Phase II trial of continuous dose-intense temozolomide in recurrent malignant glioma: RESCUE study. J Clin Oncol. 2010 Apr 20;28(12):2051-7. doi: 10.1200/JCO.2009.26.5520. Epub 2010 Mar 22. PMID 20308655
- [Background] Yung WK, Prados MD, Yaya-Tur R, Rosenfeld SS, Brada M, Friedman HS, Albright R, Olson J, Chang SM, O'Neill AM, Friedman AH, Bruner J, Yue N, Dugan M, Zaknoen S, Levin VA. Multicenter phase II trial of temozolomide in patients with anaplastic astrocytoma or anaplastic oligoastrocytoma at first relapse. Temodal Brain Tumor Group. J Clin Oncol. 1999 Sep;17(9):2762-71. doi: 10.1200/JCO.1999.17.9.2762. PMID 10561351
- [Background] Cairncross JG, Ueki K, Zlatescu MC, Lisle DK, Finkelstein DM, Hammond RR, Silver JS, Stark PC, Macdonald DR, Ino Y, Ramsay DA, Louis DN. Specific genetic predictors of chemotherapeutic response and survival in patients with anaplastic oligodendrogliomas. J Natl Cancer Inst. 1998 Oct 7;90(19):1473-9. doi: 10.1093/jnci/90.19.1473. PMID 9776413
- [Background] Van den Bent MJ, Reni M, Gatta G, Vecht C. Oligodendroglioma. Crit Rev Oncol Hematol. 2008 Jun;66(3):262-72. doi: 10.1016/j.critrevonc.2007.11.007. Epub 2008 Feb 12. PMID 18272388
- [Background] Mollemann M, Wolter M, Felsberg J, Collins VP, Reifenberger G. Frequent promoter hypermethylation and low expression of the MGMT gene in oligodendroglial tumors. Int J Cancer. 2005 Jan 20;113(3):379-85. doi: 10.1002/ijc.20575. PMID 15455350
- [Background] Gan HK, Rosenthal MA, Dowling A, Kalnins R, Algar E, Wong N, Benson A, Woods AM, Cher L. A phase II trial of primary temozolomide in patients with grade III oligodendroglial brain tumors. Neuro Oncol. 2010 May;12(5):500-7. doi: 10.1093/neuonc/nop065. Epub 2010 Feb 8. PMID 20406900